CLINICAL TRIAL: NCT04063111
Title: ROLE OF VACUUM ASSISTED CLOSURE IN OPEN TYPE III B TIBIAL FRACTURES
Brief Title: Role of Vacuum in Open Fracture Tibia Grade III Type B
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Albair Malaka Sedki, Resident of orthopedic surgery department, Assiut University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: VAC in open fracture tibia
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Open Fracture of Tibia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A (Active Comparator): Group A will be treated with vacuum assistant closure
  Interventions: Device: vacuum assistant closure
- group B (Active Comparator): Group B will be treated with conventional dressing
  Interventions: Device: CONVENTIONAL DRESSING

INTERVENTIONS:
Device: vacuum assistant closure — Expose the open wound bed to negative pressure. This pressure removes edema or hemorrhage, mechanically pulls on the wound edges, decreases in wound surface area, improves circulation, and enhances proliferation of granulation tissue that filled the soft tissue defect.
  Arms: group A
Device: CONVENTIONAL DRESSING — CONVENTIONAL DRESSING for wound of open fracture of tibia grade III B
  Arms: group B

SUMMARY:
- Evaluate the role of VAC in decreasing the time needed for soft tissue coverage and definitive fixation in open IIIB tibial fractures

DETAILED DESCRIPTION:
* Open fractures are injuries in which the skin and soft-tissue integument are disrupted and the underlying bone is exposed to the external environment. This communication results in contamination by microorganisms that can cause deep or superficial infection. Impaired vascularity, devitalized tissue, and loss of skeletal stability are all factors leading to increased susceptibility to infection after open fracture [1, 2].
* Current protocols for treating open fractures include early administration of antibiotics, timely surgical debridement, skeletal stabilization, sterile dressing, systemic support, and establishment of soft-tissue coverage in a wound environment that is clean [3, 4-8].
* VAC is being used to obviate the need for, or enhance the success of, free-flap coverage in open fractures that are significant enough to preclude primary closure, delayed primary closure, or healing by secondary intention. VAC device and its components, which in a closed system expose the open wound bed to negative pressure. This pressure removes edema or hemorrhage, mechanically pulls on the wound edges, decreases in wound surface area, improves circulation, and enhances proliferation of granulation tissue that filled the soft tissue defect, enhance debridement of wound debris, reducing the need for costly free-flap transfers. VAC devices have been used in many surgical disciplines but only recently have become popular in orthopedics [7, 9,].

ELIGIBILITY:
Inclusion Criteria:

* - Gustilo Type III B open fractures of the tibia [10].
* Skeletal mature patients.

Exclusion Criteria:

* - Bone defect more than 5 cm Gustilo Type III B open fractures of the tibia.
* Medical commodities that make the patient unfit for surgery. (e.g. Liver Cell Failure, liver cirrhosis, renal failure )

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-15 (Estimated); Primary Completion 2021-10-15 (Estimated); Study Completion 2022-04-15 (Estimated)

PRIMARY OUTCOMES:
- Time for definitive soft tissue coverage | baseline
  - Evaluate the role of VAC in decreasing the time needed for soft tissue coverage and definitive fixation in open IIIB tibial fractures

SECONDARY OUTCOMES:
- The type of soft tissue reconstruction | baseline

REFERENCES:
- [Background] Cherubino M, Valdatta L, Tos P, D'Arpa S, Troisi L, Igor P, Corradi F, Khan U. Role of Negative Pressure Therapy as Damage Control in Soft Tissue Reconstruction for Open Tibial Fractures. J Reconstr Microsurg. 2017 Oct;33(S 01):S08-S13. doi: 10.1055/s-0037-1606542. Epub 2017 Oct 6. PMID 28985633